CLINICAL TRIAL: NCT04337268
Title: Acute Effects of GLP-1 on Renal Hemodynamics: Simultaneous Perfusion and Oxygenation Measurements in Cortex and Medulla Using Magnetic Resonance Imaging
Brief Title: Acute Effects of GLP-1 on Renal Hemodynamics
Acronym: GLP1RRBF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Department of Cardiovascular and Renal Research, University of Southern Denmark (Unknown)
Responsible Party: Principal Investigator, Ali Asmar, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-18050603
Record Dates: First submitted 2020-03-29; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: The GLP-1-mediated Gut-kidney Axis
Keywords: glucagon-like peptide-1; kidney; renal hemodynamics; renal blood flow
MeSH Terms: interventions — Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- human glucagon-like peptide-1 (Active Comparator): Intervention:
  Drug: human glucagon-like peptide-1 Other names: GLP-1
  Interventions: Drug: Glucagon-Like Peptide 1
- Placebo (Placebo Comparator): Intervention:
  Drug: Placebo (saline) Other names: Placebo for human glucagon-like peptide-1
  Interventions: Drug: saline 0.9%

INTERVENTIONS:
Drug: Glucagon-Like Peptide 1 — Intravenous infusion (1.5 pmol/kg/min) for 60 min.
  Other Names: GLP-1
  Arms: human glucagon-like peptide-1
Drug: saline 0.9% — Intravenous infusion for 60 min.
  Other Names: Placebo for GLP-1
  Arms: Placebo

SUMMARY:
This study investigates the hypothesis, that GLP-1's suppression of ANG II and natriuretic action increase medullary perfusion and decrease oxygen consumption, leading to higher tissue oxygenation.

DETAILED DESCRIPTION:
Human studies have recently demonstrated a significant natriuretic effect of GLP-1 when the extracellular fluid volume (ECFV) is expanded by intravenous sodium-loading; in these studies, there was a suppression of ANG II with no change in net renal hemodynamics, pointing to a tubular mechanism for reduced NaCl reabsorption secondary to the ANG II suppression. In the current randomized and controlled study, investigators aim to test the hypothesis that GLP-1's suppression of ANG II and natriuretic action increase medullary perfusion and decrease oxygen consumption, leading to higher tissue oxygenation. Thus, contributing to the renoprotective action of GLP-1.

Under fixed sodium intake for 4 days before each study day, 10 healthy male participants will be investigated during a 1-hour infusion of GLP-1 (1.5 pmol/kg/min) or vehicle together with an intravenous infusion of 0.9% NaCl. Interleaved measurements of RAF, oxygenation (T2*) and perfusion by arterial spin labeling in the renal cortex and medulla at fixed time points will be conducted, using Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Normal health demonstrated by medical examination.
* Normal values for fasting plasma glucose, total cholesterol, triglyceride, HDL, LDL, creatinine, AST, ALT and electrolyte concentrations.

Exclusion Criteria:

* Immunosuppressive treatment for the previous 12 months.
* Alcohol abuse.
* Medical treatment with oral glucocorticoids, dipeptidyl peptidase-4 (DPP-4) inhibitors, or GLP-1 receptor agonists that, in the opinion of the investigator, may interfere with glucose metabolism.
* Use of lithium.
* Medical treatment that affects insulin secretion or cardiovascular efficacy goals.
* Liver disease (ALT> 2 x normal value).
* Renal impairment (creatinine> 130 µM and / or albuminuria).
* Severe claustrophobia.
* MRI incompatible foreign bodies.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
T2* signal | 1 hour
  Changes in T2* signal in renal cortex and medulla
Arterial Spin Labeled (ASL) | 1 hour
  Changes in Arterial Spin Labeled (ASL) MRI Perfusion Imaging in renal cortex and medulla
Renal Artery Flow Phase (RAF) | 1 hour
  Changes in Renal Artery Flow Phase (RAF)-Contrast Magnetic Resonance

CONTACTS AND LOCATIONS:
Overall Officials: Ali Asmar, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet - Glostrup, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holst JJ. The physiology of glucagon-like peptide 1. Physiol Rev. 2007 Oct;87(4):1409-39. doi: 10.1152/physrev.00034.2006. PMID 17928588
- [Background] Korner M, Stockli M, Waser B, Reubi JC. GLP-1 receptor expression in human tumors and human normal tissues: potential for in vivo targeting. J Nucl Med. 2007 May;48(5):736-43. doi: 10.2967/jnumed.106.038679. PMID 17475961
- [Background] Pyke C, Heller RS, Kirk RK, Orskov C, Reedtz-Runge S, Kaastrup P, Hvelplund A, Bardram L, Calatayud D, Knudsen LB. GLP-1 receptor localization in monkey and human tissue: novel distribution revealed with extensively validated monoclonal antibody. Endocrinology. 2014 Apr;155(4):1280-90. doi: 10.1210/en.2013-1934. Epub 2014 Jan 27. PMID 24467746
- [Background] Asmar A, Simonsen L, Asmar M, Madsbad S, Holst JJ, Frandsen E, Moro C, Jonassen T, Bulow J. Renal extraction and acute effects of glucagon-like peptide-1 on central and renal hemodynamics in healthy men. Am J Physiol Endocrinol Metab. 2015 Apr 15;308(8):E641-9. doi: 10.1152/ajpendo.00429.2014. Epub 2015 Feb 10. PMID 25670826
- [Background] Asmar A, Simonsen L, Asmar M, Madsbad S, Holst JJ, Frandsen E, Moro C, Sorensen CM, Jonassen T, Bulow J. Glucagon-like peptide-1 does not have acute effects on central or renal hemodynamics in patients with type 2 diabetes without nephropathy. Am J Physiol Endocrinol Metab. 2016 May 1;310(9):E744-53. doi: 10.1152/ajpendo.00518.2015. Epub 2016 Mar 8. PMID 26956188
- [Background] Asmar A, Asmar M, Simonsen L, Madsbad S, Holst JJ, Hartmann B, Sorensen CM, Bulow J. Glucagon-like peptide-1 elicits vasodilation in adipose tissue and skeletal muscle in healthy men. Physiol Rep. 2017 Feb;5(3):e13073. doi: 10.14814/phy2.13073. PMID 28174344
- [Background] Skov J, Dejgaard A, Frokiaer J, Holst JJ, Jonassen T, Rittig S, Christiansen JS. Glucagon-like peptide-1 (GLP-1): effect on kidney hemodynamics and renin-angiotensin-aldosterone system in healthy men. J Clin Endocrinol Metab. 2013 Apr;98(4):E664-71. doi: 10.1210/jc.2012-3855. Epub 2013 Mar 5. PMID 23463656
- [Background] Asmar A, Cramon PK, Simonsen L, Asmar M, Sorensen CM, Madsbad S, Moro C, Hartmann B, Jensen BL, Holst JJ, Bulow J. Extracellular Fluid Volume Expansion Uncovers a Natriuretic Action of GLP-1: A Functional GLP-1-Renal Axis in Man. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2509-2519. doi: 10.1210/jc.2019-00004. PMID 30835273
- [Derived] Haddock B, Kristensen KB, Tayyab M, Larsson HBW, Lindberg U, Vestergaard M, Francis S, Jensen BL, Andersen UB, Asmar A. GLP-1 Promotes Cortical and Medullary Perfusion in the Human Kidney and Maintains Renal Oxygenation During NaCl Loading. J Am Heart Assoc. 2023 Feb 7;12(3):e027712. doi: 10.1161/JAHA.122.027712. Epub 2023 Feb 3. PMID 36734354